CLINICAL TRIAL: NCT03116841
Title: Vonoprazan Study of Investigating the Effect on Sleep Disturbance Associated With Reflux Esophagitis- Exploratory Evaluation (VISTAEXE)
Brief Title: Vonoprazan Study of Investigating the Effect on Sleep Disturbance Associated With Reflux Esophagitis- Exploratory Evaluation
Acronym: VISTAEXE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vonoprazan-4006; U1111-1192-9760 (Registry Identifier: WHO); JapicCTI-173538 (Registry Identifier: Japic-CTI)
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Reflux Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vonoprazan 20 mg (Experimental): Vonoprazan 20 mg orally administered once daily
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan 20 mg

SUMMARY:
The purpose of this study is to exploratorily evaluate the effect of vonoprazan 20 mg on sleep disturbance of patients with reflux esophagitis, who have heartburn and/or regurgitation and ≥ 6.0 in the Pittsburgh Sleep Quality Index (PSQI) global score despite the maintenance treatment with PPI other than vonoprazan.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of vonoprazan on sleep disturbance in the participants under maintenance treatment for reflux esophagitis with proton pump inhibitor (PPI) other than vonoprazan after initial treatment.

Participants who have been diagnosed as reflux esophagitis based on Los Angeles (LA) Classification Grades A to D, undergoing maintenance treatment with PPI other than vonoprazan after initial treatment, and with Pittsburgh Sleep Quality Index (PSQI) global score >= 6.0 at enrolment (VISIT 1) will be eligible for study entry and will be administered vonoprazan 20 mg once daily for 8 weeks.

Planned number of participants is 25. The study period is 9 weeks. The number of visits is 6visits.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who completed the initial treatment with PPIs (esomeprazole, omeprazole, rabeprazole, or lansoprazole) and have received high dose PPIs (esomeprazole 20 mg, omeprazole 20 mg, rabeprazole 10 mg, or lansoprazole 30 mg) for more than 8 weeks at the time of informed consent as maintenance treatment for LA Classification Grades A to D reflux esophagitis.
2. Participants who have heartburn and/or regurgitation.
3. Participants with reflux esophagitis related sleep disturbance, fulfilling at least one of following in a week before the baseline/start of administration.

   * Difficulty in falling asleep for > = 3 nights
   * Nocturnal awaking or early morning awaking for > = 3 nights
4. Participants whose heartburn and/or regurgitation at the time of informed consent were alleviated from initial treatment.
5. Participants with PSQI global score > = 6.0
6. Participants who, in the opinion of the investigator, are capable of understanding the content of the study and complying with the protocol requirements.
7. Participants who can sign and date an informed consent form and information sheet prior to the initiation of the study procedures.
8. Male or female participants aged 20 years or older at the time of informed consent.
9. Therapeutic category: Ambulatory

Exclusion Criteria:

1. Participants with Zollinger-Ellison syndrome.
2. Participants with diseases that affect sleep (chronic obstructive pulmonary disease, bronchitis asthma, sleep apnea syndrome, mental disorder, etc.)
3. Nightshift workers.
4. Participants who have a plan to travel beyond three time zones during the study.
5. Participants with a history of, concurrent, or suspicious functional dyspepsia or functional heartburn based on Rome IV criteria.
6. Participants with history of surgery or treatment affecting gastroesophageal reflux (fundoplication or dilation for esophageal stenosis [except for Schatzki's ring], etc.).
7. Participants with an esophagus-related complication (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal stenosis, etc.), a history of radiotherapy or cryotherapy of the esophagus, a caustic or physiochemical trauma (esophageal sclerotherapy, etc.). However, participants with Schatzki's ring (mucosal tissue ring around inferior esophageal sphincter) or Barrett's esophagus are allowed to be included.
8. Participants with a history of gastrectomy, gastrointestinal resection, or vagotomy.
9. Participants who took antidepressant agents or anti-anxiety agents within 8 weeks before the time of informed consent.
10. Participants who took H2 receptor antagonist within 8 weeks before the time of informed consent.
11. Participants planning to take prohibited concomitant medications during the study period.
12. Participants who have any of the following abnormal clinical laboratory test values at the screening (VISIT 1):

    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN)
    * Bilirubin (Total bilirubin) > ULN
13. Participants with a malignant tumor.
14. Participants who are pregnant, breast-feeding, possibly pregnant, or planning to become pregnant.
15. Participants who have serious renal diseases.
16. Participants with the conditions listed under administration contraindication in the vonoprazan package insert.
17. Participants participating in other clinical studies.
18. Participants who have been determined as inappropriate participants by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- Japan (6):
  - Tokatsu Tsujinaka Hospital, Abiko, Chiba
  - Amada Clinic, Kōriyama, Fukushima
  - Aoyama Clinic, Kobe, Hyōgo
  - Kashiwara Municipal Hospital, Kashihara, Osaka
  - Saino Clinic, Tokorozawa, Saitama
  - Masuyama Clinic, Ōtawara, Tochigi

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study in Japan, from 02 August 2017 to 20 December 2017.
Pre-assignment Details: Participants with a historical diagnosis of reflux esophagitis, undergoing maintenance treatment with a proton pump inhibitors (PPI) after initial treatment, and with Pittsburgh Sleep Quality Index (PSQI) global score ≥ 6.0 at the start of administration (VISIT 2) were enrolled and was administered vonoprazan 20 mg once daily for 8 weeks.
Groups:
- Vonoprazan 20mg: Vonoprazan 20 mg, orally, once daily, for up to 8 weeks.
Period: Overall Study
Arm/Group | Vonoprazan 20mg
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Age, Customized [Number; unit: Participants]
  >=20 and <80 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes From Start of Administration (Week 0) in Pittsburgh Sleep Quality Index (PSQI) Global Score at End of Study
Description: PSQI is a self-rated questionnaire for sleep quality. It includes 18 items across 7 components; C1: Sleep quality, C2: Sleep latency, C3: Sleep duration, C4: Sleep efficiency, C5: Sleep disturbance, C6: Use of sleep medication, C7: Daytime dysfunction. Each component is scored 0-3 (0 = no difficulty, 3=severe difficulty), and total score ranging from 0 to 21. Higher scores are representing worse sleep quality. Reported data were individual scores for each participant (Participant A to C) since descriptive statistics value was not calculated due to small size population (totally 3 participants).
Time Frame: Week 0 to End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Scores on a Scale
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Scores on a Scale
  Participant A: number analyzed (Participants) | 1
  Participant A | -2
  Participant B: number analyzed (Participants) | 1
  Participant B | 1
  Participant C: number analyzed (Participants) | 1
  Participant C | -6

2. Secondary Outcome: Changes From Start of Administration (Week 0) in PSQI Global Score at Week 4
Description: PSQI is a self-rated questionnaire for sleep quality. It includes 18 items across 7 components; C1: Sleep quality, C2: Sleep latency, C3: Sleep duration, C4: Sleep efficiency, C5: Sleep disturbance, C6: Use of sleep medication, C7: Daytime dysfunction. Each component is scored 0-3 (0 = no difficulty, 3=severe difficulty), and total score ranging from 0 to 21. Higher scores are representing worse sleep quality. Reported data were individual scores for each participants (Participant A to C) since descriptive statistics value was not calculated due to small size population (totally 3 participants).
Time Frame: From Week 0 to Week 4
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Scores on a Scale
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Scores on a Scale
  Participant A: number analyzed (Participants) | 1
  Participant A | -2
  Participant B: number analyzed (Participants) | 1
  Participant B | 1
  Participant C: number analyzed (Participants) | 1
  Participant C | -5

3. Secondary Outcome: Percentage of Participants With PSQI Global Score <6.0 at Week 4 and End of Study
Description: PSQI is a self-rated questionnaire for sleep quality. It includes 18 items across 7 components; C1: Sleep quality, C2: Sleep latency, C3: Sleep duration, C4: Sleep efficiency, C5: Sleep disturbance, C6: Use of sleep medication, C7: Daytime dysfunction. Each component is scored 0-3 (0 = no difficulty, 3=severe difficulty), and total score ranging from 0 to 21. Higher scores are representing worse sleep quality.
Time Frame: Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Percentage of Participants
  Week 4 | 33.3
  End of study | 66.7

4. Secondary Outcome: Changes From Start of Administration (Week 0) in C1: Sleep Quality of PSQI Global Score at Week 4 and End of Study
Description: as for outcome 2
Time Frame: Week 0, Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Scores on a Scale
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Scores on a Scale
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | 0
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | -1
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | 0
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 0
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | -2
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | -2

5. Secondary Outcome: Changes From Start of Administration (Week 0) in C2: Sleep Latency of PSQI Global Score at Week 4 and End of Study
Description: as for outcome 2
Time Frame: Week 0, Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Scores on a Scale
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Scores on a Scale
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | -1
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | -1
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | 0
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 0
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | -1
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | -1

6. Secondary Outcome: Changes From Start of Administration (Week 0) in C3: Sleep Duration of PSQI Global Score at Week 4 and End of Study
Description: as for outcome 2
Time Frame: Week 0, Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Scores on a Scale
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Scores on a Scale
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | 0
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | 0
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | 1
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 1
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | 0
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | -1

7. Secondary Outcome: Changes From Start of Administration (Week 0) in C4: Sleep Efficiency of PSQI Global Score at Week 4 and End of Study
Description: as for outcome 2
Time Frame: Week 0, Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Scores on a Scale
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Scores on a Scale
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | 0
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | 0
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | 0
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 0
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | 0
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | 0

8. Secondary Outcome: Changes From Start of Administration (Week 0) in C5: Sleep Disturbance of PSQI Global Score at Week 4 and End of Study
Description: as for outcome 2
Time Frame: Week 0, Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Scores on a Scale
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Scores on a Scale
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | 0
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | 0
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | 0
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 0
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | 0
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | 0

9. Secondary Outcome: Changes From Start of Administration (Week 0) in C7: Daytime Dysfunction of PSQI Global Score at Week 4 and End of Study
Description: as for outcome 2
Time Frame: Week 0, Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Scores on a Scale
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Scores on a Scale
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | -1
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | 0
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | 0
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 0
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | -2
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | -2

10. Secondary Outcome: Number of Nocturnal Awakenings Assessed by a Question at Week 4, and End of Study
Description: Number of nocturnal awakenings was assessed by a question about nocturnal awakenings, "How Many Times Wake Up?" which was asked to each participants by investigator. Reported data were individual times for each participants (Participant A to C) since descriptive statistics value was not calculated due to small size population (totally 3 participants).
Time Frame: Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Nocturnal awakenings
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Nocturnal awakenings
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | 0
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | 0
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | 1
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 2
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | 1
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | 1

11. Secondary Outcome: Percent Changes From Start of Administration (Week 0) in Actigraph-Measured Sleep Efficiency at Week 4, and End of Study
Description: Actigraph is a small device usually that records the activity level of the body by sensing physical movement and that is used especially to measure the amount and quality of sleep. Mean value from the past 7 days at each time point was used for calculation. Reported data were individual values for each participants (Participant A to C) since descriptive statistics value was not calculated due to small size population (totally 3 participants).
Time Frame: Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Percent of Change
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Percent of Change
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | 3.10
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | 4.48
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | -10.56
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 3.57
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | 2.00
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | -3.17

12. Secondary Outcome: Changes From Start of Administration (Week 0) in Actigraph-Measured Sleep Latency at Week 4, and End of Study
Description: Actigraph is a small device usually that records the activity level of the body by sensing physical movement and that is used especially to measure the amount and quality of sleep. Reported data were individual values for each participants (Participant A to C) since descriptive statistics value was not calculated due to small size population (totally 3 participants).
Time Frame: Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Minutes
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Minutes
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | -10.00
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | -5.00
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | 21.00
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | 10.00
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | -13.00
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | 1.00

13. Secondary Outcome: Changes From Start of Administration (Week 0) in Actigraph-Measured Number of Nocturnal Awakenings at Week 4, and End of Study
Description: Actigraph is a small device usually that records the activity level of the body by sensing physical movement and that is used especially to measure the amount and quality of sleep. Mean value from the past 7 days at each time point was used for calculation. Reported data were individual times for each participants (Participant A to C) since descriptive statistics value was not calculated due to small size population (totally 3 participants).
Time Frame: Week 4 and End of study (up to Week 8)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: Nocturnal awakenings
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Nocturnal awakenings
  Participant A - Week 4: number analyzed (Participants) | 1
  Participant A - Week 4 | 0.15
  Participant A - End of study: number analyzed (Participants) | 1
  Participant A - End of study | 0.00
  Participant B - Week 4: number analyzed (Participants) | 1
  Participant B - Week 4 | -2.00
  Participant B - End of study: number analyzed (Participants) | 1
  Participant B - End of study | -1.15
  Participant C - Week 4: number analyzed (Participants) | 1
  Participant C - Week 4 | 0.86
  Participant C - End of study: number analyzed (Participants) | 1
  Participant C - End of study | 1.00

14. Secondary Outcome: Number of Participants Reporting Who Had One or More Treatment-emergent Adverse Event (TEAE)
Time Frame: Up to Week 8
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 20mg
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to Week 8
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vonoprazan 20mg
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 20mg (N=3)
Viral upper respiratory tract (Infections and infestations) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03116841/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03116841/SAP_001.pdf